CLINICAL TRIAL: NCT01581619
Title: A Phase I Study of Once-Daily External-Beam Partial-Breast Irradiation (PBI) for Selected Patients With Early Invasive N0 or Non-Invasive Breast Cancer
Brief Title: External-Beam Partial-Breast Irradiation for Early Breast Cancer 40 Gy QD Over 2 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Alphonse Taghian, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-351
Record Dates: First submitted 2012-01-11; First posted 2012-04-20 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
Keywords: Early Invasive N0; Non-Invasive
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Partial Breast Irradiation (Experimental): Partial Breast Irradiation using 40 Gy in 10 fractions over 2 weeks
  Interventions: Radiation: External Beam Partial-Breast Irradiation

INTERVENTIONS:
Radiation: External Beam Partial-Breast Irradiation — 40 Gy in ten daily fractions over two weeks

SUMMARY:
Standard therapy for patients with early stage breast cancer consists of surgery to remove the cancer followed by radiation therapy. One question regarding radiation therapy for early stage breast cancer is whether the entire breast needs to be radiated or only a more limited area surrounding the tumor. Whole-breast irradiation (WBI) is radiation therapy given to the whole breast. Partial-breast irradiation (PBI) is radiation therapy given only to the area of the breast where the cancer was removed (called the "tumor bed").

The investigators hope the option of PBI will reduce side effects from radiation therapy and shorten the radiation treatment process when compared to WBI, since only part of the breast is being treated. The investigators also hope that this will make such treatment more convenient for breast cancer patients.

The purpose of the study is to evaluate the the safety of external-beam PBI in selected early breast cancer patients utilizing PBI in ten daily fractions over two weeks. The investigators will also evaluate the local control and the cosmetic results.

DETAILED DESCRIPTION:
After signing the consent form, the following will be assessed.

-CT scan of the breast that had the cancer removed to help plan the radiation therapy. This is referred to as a CT-simulation. This scan is done routinely as part of the regular treatment.

PBI Study Treatment: You will be given PBI once daily over 10 treatment days (Mon-Fri) over a 2 week period. During this time you will have a weekly interview, physical examination, and your skin will be assessed for any side effects of the radiation.

PBI will begin between 4 weeks to 3 months after breast surgery or 2-6 weeks after chemotherapy (if you have been given chemotherapy).

After the final dose of the study:

You will have the following scheduled follow-up visits: one at the completion of the radiation, once or twice during weeks 3-9 after the completion of radiation, once every 6 months for five years, and then once every year for the following five years after the completion of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Unicentric Stage I invasive ductal breast cancer or Grade I or II DCIS measuring less than or equal to 2cm on pathology and/or mammography
* Histologically negative tumor margin 2 mm or more from any inked edges, or no tumor in a re-excision specimen or final shaved specimen
* Clips must be placed in the lumpectomy cavity at the time of final excision in order to aid in the delineation of the tumor cavity at the time of simulation and radiation delivery

Exclusion Criteria:

* No distant metastasis
* Not pregnant or breastfeeding
* No diffuse suspicious microcalcifications
* No prior radiation therapy to the ipsilateral or contralateral breast or thorax
* No histologic evidence of lymphovascular invasion (LVI)
* No histologic evidence of EIC
* No history of cosmetic or reconstructive breast surgery
* No psychiatric illness that would prevent the patient from giving informed consent
* No medical conditions that, in the opinion of the treating physician would make this protocol unreasonably hazardous for the patient
* No other currently active second malignancy other than non-melanoma skin cancers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-05; Primary Completion 2016-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Beth Isreal Deaconness Medical Center, Boston, Massachusetts
  - Brigham and Women's Hosptial, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Partial Breast Irradiation
Started | 54
Completed | 52
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Partial Breast Irradiation
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 51
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54
Method of Initial Diagnosis [Count of Participants; unit: Participants] — Population: The participant that withdrew consent was not included in the analysis
  Participants
    Mammogram: number analyzed (Participants) | 53
    Mammogram | 51
    MRI ( magnetic resonance imaging): number analyzed (Participants) | 53
    MRI ( magnetic resonance imaging) | 1
    Other: number analyzed (Participants) | 53
    Other | 1
Side of the breast cancer [Count of Participants; unit: Participants] — Population: Participant that withdrew consent was not included
  Participants
    Left Breast: number analyzed (Participants) | 53
    Left Breast | 27
    Right Breast: number analyzed (Participants) | 53
    Right Breast | 26
Stage [Count of Participants; unit: Participants] — Breast Cancer Staging:
  * Stage 0: No tumor in lymph nodes; Carcinoma in situ: with cancer cells within lobules and ducts only (no invasion)
  * Stage 1: Small invasive tumor that has not spread to the lymph nodes Population: Participant that withdrew consent was not included
  Participants
    Stage 0: number analyzed (Participants) | 53
    Stage 0 | 8
    Stage 1: number analyzed (Participants) | 53
    Stage 1 | 45
T staging [Count of Participants; unit: Participants] — T staging uses T plus a number (0 to 4) to describe the size and location of the tumor
  * Tis: Refers to carcinoma in situ, meaning the cancer is confined within the lobules or ducts of the breast tissue and has not spread into the surrounding tissue of the breast.
  * T1: The invasive part of the tumor is less than or equal to 20 millimeters (mm) at its widest diameter. T1 is further broken down to 3 sub-stages by size (a-c)
    * T1a: Tumor is larger than 1mm, but 5 mm or smaller
    * T1b: Tumor is larger than 5mm, but 10 mm or smaller
    * T1c: Tumor is larger than 10mm, but 20 mm or smaller Population: Participant that withdrew consent is not included
  Participants
    Tis: number analyzed (Participants) | 53
    Tis | 8
    T1a: number analyzed (Participants) | 53
    T1a | 17
    T1b: number analyzed (Participants) | 53
    T1b | 22
    T1c: number analyzed (Participants) | 53
    T1c | 6
Her2 FISH [Count of Participants; unit: Participants] — FISH (Fluorescence In Situ Hybridization) test for expression of Her2 (human epidermal growth factor receptor 2). Positive results indicate that Her2 is being expressed while negative indicates that Her2 is not expressed. Population: The participant that withdrew consent was not included in the analysis
  Participants
    Negative: number analyzed (Participants) | 53
    Negative | 40
    Positive: number analyzed (Participants) | 53
    Positive | 1
    Not Done: number analyzed (Participants) | 53
    Not Done | 12
Her2 IHC [Count of Participants; unit: Participants] — Immunohistochemistry (IHC) test to show if the tumor cells have Her2 receptors on their surface. IHC test gives a score from 0 to 3+ that measures the amount of Her2 receptor protein on the surface of the cancer cells. A score of either 0 or 1+ is considered Her2 negative, a score of 2+ is considered borderline, a score of 3+ is considered positive. The positive result means that the cells are expressing the Her2 protein. Population: The participant that withdrew consent was not included in the analysis
  Participants
    (3+) / Her2 Positive: number analyzed (Participants) | 53
    (3+) / Her2 Positive | 1
    (2+) / Borderline: number analyzed (Participants) | 53
    (2+) / Borderline | 4
    (0, 1+) Her2 Negative: number analyzed (Participants) | 53
    (0, 1+) Her2 Negative | 34
    Not Done: number analyzed (Participants) | 53
    Not Done | 14
Estrogen Receptor [Count of Participants; unit: Participants] — Test whether the cancer cells express estrogen receptors.
  * Positive: Estrogen receptors detected
  * Negative: Estrogen receptors not detected Population: The participant that withdrew consent was not included in the analysis
  Participants
    Positive: number analyzed (Participants) | 53
    Positive | 53
    Negative: number analyzed (Participants) | 53
    Negative | 0
Progesterone Receptor [Count of Participants; unit: Participants] — Test for the presence of Progesterone receptors on the cancer cells. Positive indicates that they are present, Few/ faint cells indicates a borderline result, negative indicates they were not detected. Population: The participant that withdrew consent was not included in the analysis
  Participants
    Positive: number analyzed (Participants) | 53
    Positive | 47
    Few/ Faint Cells: number analyzed (Participants) | 53
    Few/ Faint Cells | 3
    Negative: number analyzed (Participants) | 53
    Negative | 3
Histologic Grade [Count of Participants; unit: Participants] — Differentiation refers to how similar cancer tissue is to normal tissue. Well differentiated cancer tissue looks more like normal tissue and tends to grow or spread more slowly than poorly differentiated cancer tissue which looks less like normal tissue. Population: The participant that withdrew consent was not include in the analysis
  Participants
    Well Differentiated: number analyzed (Participants) | 53
    Well Differentiated | 21
    Moderately Differentiated: number analyzed (Participants) | 53
    Moderately Differentiated | 26
    Poorly Differentiated: number analyzed (Participants) | 53
    Poorly Differentiated | 1
    Other: number analyzed (Participants) | 53
    Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety of External-beam PBI Utilizing 40Gy in Ten Daily Fractions Over Two Weeks
Description: The safety of external-beam PBI in selected stages 0 and I female breast cancer patients utilizing 40 Gy in ten daily fractions over two weeks. The study will be deemed too toxic if >10% of enrolled patients have at least one of the following outcomes within 24 months of completion of PBI.
  1. Grade 3 or 4 skin/subcutaneous or pulmonary toxicity.
  2. The development of clinical fat necrosis.
  3. The development of rib fracture on the ipsilateral treated side, detected either clinically and/or radiographically.
  The data is shown as the number of participants that experienced each of the specific toxicities.
Time Frame: 2 years
Population: Analysis does not include the one participant who withdrew consent before outcome was met.
Measure: Count of Participants; unit: Participants
Arm/Group | Partial Breast Irradiation
Number analyzed (Participants) | 53
Participants
  Grade 3 or 4 Skin/ Subcutaneous toxicity | 0
  Grade 3 or 4 Pulmonary Toxicity | 0
  Fat Necrosis | 0
  Rib fractures on ipsilateral treated side | 0

2. Secondary Outcome: Local Control Rates
Description: The local control rates (analyzed separately for patients with DCIS and invasive cancer). Local control is defined as lack of recurrence in the treated breast and ipsilateral axillary, supraclavicular and internal mammary lymph nodes. Recurrence is defined as the regrowth of tumor cells left following initial therapy and/or the development of new primary tumors unrelated to the original one. DCIS stands for 'Ductal Carcinoma In Situ'.
Time Frame: 2 years
Population: The one participant that withdrew consent before the outcome was met was excluded from the analysis
Measure: Count of Participants; unit: Participants
Groups:
- Partial Breast Irradiation - DCIS Only: Partial Breast Irradiation using 40 Gy in 10 fractions over 2 weeks
  External Beam Partial-Breast Irradiation: 40 Gy in ten daily fractions over two weeks
  Participants with DCIS only
- Partial Breast Irradiation - Invasive Cancer: Partial Breast Irradiation using 40 Gy in 10 fractions over 2 weeks
  External Beam Partial-Breast Irradiation: 40 Gy in ten daily fractions over two weeks
  Participants with Invasive breast cancer
Arm/Group | Partial Breast Irradiation - DCIS Only | Partial Breast Irradiation - Invasive Cancer
Number analyzed (Participants) | 8 | 45
Participants
  Local Control | 8 | 45
  Local Recurrence | 0 | 0

3. Secondary Outcome: Distant Control Rates
Description: The number of participants that achieved distant control. Distant control is defined as a lack of distant metastasis following the completion of treatment. Distant metastasis refers to the development of disease at distant body sites like the lung, liver, bone, or brain.
Time Frame: 2 years
Population: The one participant that withdrew consent before the outcome was met was excluded from the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Partial Breast Irradiation
Number analyzed (Participants) | 53
Participants
  Distant Control | 53
  Distant Metastasis | 0

4. Secondary Outcome: Breast Cosmesis
Description: Breast Cosmesis was assessed using a cosmetic scoring system. The data shown represent the latest assessment for each participant at the time of analysis. Cosmetic changes were assessed using the following the following criteria.
  * Excellent: Little or no observable change
  * Good: Minimal but identifiable changes
  * Fair: Significant results of radiotherapy noted
  * Poor: Severe normal tissue sequelae
Time Frame: End of treatment, 4-9 weeks post treatment, every six months for first 5 years, then annually for 5 years
Population: The one participant that withdrew consent before outcomes were met was excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Partial Breast Irradiation
Number analyzed (Participants) | 53
Participants
  Excellent | 39
  Good | 12
  Fair | 2
  Poor | 0

ADVERSE EVENTS:
Time Frame: Toxicity is assessed at the end of treatment (two weeks), once or twice at 3-9 weeks post treatment, then every six months for 5 years, then once every year for five fear (total of 10 years). Median duration of 28 months at the time of analysis.
Description: The participant that withdrew consent was not able to be assessed for adverse events and was not included in the adverse event analysis.
Arm/Group | Partial Breast Irradiation
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 2/53
Other Adverse Events (participants affected / at risk) | 47/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Partial Breast Irradiation (N=53)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1) — Cellulitis
Seroma (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Partial Breast Irradiation (N=53)
Breast pain (Reproductive system and breast disorders) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 34 (41)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5 (6)
Fatigue (General disorders) | 19 (19)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 8 (9)
Hot flashes (Vascular disorders) | 1 (1)
Localized edema (General disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 27 (31)
Skin induration (Skin and subcutaneous tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes